CLINICAL TRIAL: NCT01565447
Title: Temporal and Spatial Gait Parameters of Children Undergoing Treatment for and Surviving Acute Lymphoblastic Leukemia and Lymphoblastic Lymphoma
Brief Title: Acute Lymphoblastic Leukemia (ALL) and Lymphoblastic Lymphoma Gait Parameters Study
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Nancy Durben, Assistant Professor of Physical Therapy, Oregon Health and Science University
Other Study IDs: OregonHSU
Record Dates: First submitted 2012-01-31; First posted 2012-03-28 (Estimated); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Acute Lymphoblastic Leukemia; Childhood Lymphoblastic Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Children with ALL or LL: Children diagnosed with ALL or LL will be recruited for this study

SUMMARY:
This purpose of this study it to characterize the walking patterns of children diagnosed with Acute Lymphoblastic Leukemia (ALL)and Lymphoblastic Lymphoma (LL) at different times in the treatment protocol and after completion of treatment. Their walking patterns will be compared to children without ALL or LL to see if their walking patterns are different at specific times in their treatment program or up to 10 years after completion of their treatment. The investigators will gather data by observing how the child walks, runs, hops on one foot and climbs stairs and by recording walking patterns on a pressure sensitive mat. The investigators will compare this data to children without ALL and LL.

DETAILED DESCRIPTION:
Cases will be identified and referred by the primary oncologist or by the Childhood Cancer Survivorship team. When a possible subject has been identified they will be contacted via telephone or during a routine clinic visit to determine their interest in the study. Two hundred subjects will be recruited for participation with the goal of 5-10 subjects at each of the 14 times points across the treatment protocol and survivorship. These time points to include: at diagnosis, the start of consolidation therapy, the start of interim maintenance therapy, the start of delayed intensification therapy, Day 29 of delayed intensification therapy, the start of interim maintenance II therapy (if applicable), Day 1 of cycle 1,3,5 of maintenance therapy, end of therapy, and 1, 3, 5, and 10 years off therapy ( +/-1 year).

Clinical data will be collected from the medical record, roadmaps documenting cancer-directed therapy, direct patient interview and examination by the physical therapist during the study evaluation. Clinical data will include: Date of birth (to calculate age at diagnosis and current age); Gender; Race and Ethnicity; Primary cancer diagnosis; Date of Primary Cancer Diagnosis; Chemotherapeutic agents received (agent name, cumulative dose and date received); Radiation therapy (date received, site radiated, and dose delivered); Any other clinical conditions affecting musculoskeletal performance; Dates of previous PT; Pain score at the time of study participation. Height, weight, shoe size and leg length will be collected at time of study participation.

Subjects will complete a self report of the PedsQL™ Generic Core Scale and the parents will complete the parental report.

Observation gait assessment will include hopping on one foot, running and walking 30' and ascending/descending stairs.

Temporal spatial gait parameters will be recorded on the GaitRite mat

ELIGIBILITY:
Inclusion Criteria:

1. Age 2-27 years of age
2. Diagnosis of acute lymphoblastic leukemia or lymphoblastic lymphoma
3. Currently undergoing treatment for ALL or LL or completed treatment for ALL or LL in the last 10 years.

Exclusion Criteria

1. Relapsed ALL or LL
2. Received a stem cell transplant, either autologous or allogeneic
3. Non ambulatory status prior to diagnosis of acute lymphoblastic leukemia or lymphoblastic lymphoma

Ages: 2 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children diagnosed with ALL or LL and are currently undergoing treatment for or have survived treatment and are no more than 10 years post completion of treatment
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
Temporal and Spatial Gait | At diagnosis, start of consolidation tx, the start of interim maintenance tx, the start of delayed intensification tx, Day 29 of delayed intensification tx, the start of interim maintenance II tx (if applicable), Day 1 of cycle, 1,3,5 of maintenance tx.
  To characterize temporal and spatial gait parameters of children with ALL/LL at specific time points during their treatment and survivorship using the GAITRite® evaluation system.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Lindemulde, MD, MCR, Study Director — Oregon Health and Science University
Locations (1):
- Doernbecher Children Hospital, Portland, Oregon, United States